CLINICAL TRIAL: NCT06697899
Title: Food Effect on Pharmacokinetic Profile for TGRX-678 Tablet in Chinese Healthy Subject With Single Oral Administration
Brief Title: TGRX-678 Phase I Oral Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen TargetRx, Inc. (Industry)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TGRX-678-1002
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fasting (Experimental): Participants take TGRX-678 under fasting state
  Interventions: Drug: TGRX-678
- Low-fat Diet (Experimental): Participants take TGRX-678 after low-fat meal intake
  Interventions: Drug: TGRX-678
- High-fat Diet (Experimental): Participants take TGRX-678 after high-fat meal intake
  Interventions: Drug: TGRX-678

INTERVENTIONS:
Drug: TGRX-678 — All participants are given TGRX-678 orally at 240 mg

SUMMARY:
A study evaluating the effects of food intake on the pharmacokinetic (PK) profiles of TGRX-678

DETAILED DESCRIPTION:
This study is designed as single-center, single-dose, randomized, open-label and parallel-comparison to evaluate food effect on PK profile of TGRX-678 in healthy subjects. Safety and tolerability of the drug is also evaluated during study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants, male or female
* Age between 18 and 45 (both inclusive)
* Body Weight: male ≥ 50 kg, female ≥ 45 kg; Body Mass Index (BMI) between 19.0 and 26.0 kg/m^2 (both inclusive)
* Signing informed concent at own will
* Able to communicate with researcher and able to complete study per protocol instruction

Exclusion Criteria:

* Clinically significant abnormal results in lab test, physical exam or 12-lead electrocardiogram (ECG) test
* Positive results for Hepatitis B, Hepatitis C, HIV or Syphilis
* QT interval elongation as indicated by 12-lead ECG test during screening period
* Use of any medication that could impact CYP3A4 enzyme activities within 30 days prior to Screening period
* Use of any medication within 14 days of first dose of the investigational drug
* Vaccinated within 30 days of first dose of the investigational drug, or planning to be vaccinated during study
* History of instrumental cardiovascular diseases
* Received major surgery within 6 months prior to Screening, or with surgical wounds not completely healed
* History of any severe disease or conditions that could affect study results per investigator's discretion
* History of allergic conditions or is allergic to components of the investigational drug
* Having conditions that could affect drug absorption or difficulties to swallow
* History of smoking of >5 cigarettes per day within 3 months prior to screening, or cannot stop tabacco using during study
* History of alcohol abuse, or alcohol consumption of >14 unit alcohol within 3 months prior to screening
* History of substance use, or tested positive for drug test during screening
* History of specific food (i.e., grapefruit, mango) consumption, or/and large tea/coffee/caffeinated drink/grapefruit product intake of > 8 cups per day, within 2 weeks prior to first dose
* Having special dietary requirement and cannot comply with food requirement of the study
* Pregnant or breastfeeding female, or tested positive in pregnancy test
* History of unprotected sexual activities within 1 month prior to screening
* Having plans for pregnancy during the study and within 6 months after study completion; or not agreeing to take strict contraceptive measures during study and within 6 months after study completion
* History of blood loss/ blood donation of ≥ 400 mL within 3 months prior to screening, or planning to donate blood within 1 month after study completion
* Any reasons that is deemed unsuitable for study participation as determined by investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2024-11-24 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Plasma Tmax | During Treatment period (Day 1 to Day 43)
  Time to maximum concentration (Tmax) of TGRX-678 measured in plasma
Plasma Tlag | During Treatment period (Day 1 to Day 43)
  Time between drug administration to drug absorption (Tlag) as indicated by TGRX-678 plasma concentration
Plasma Cmax | During Treatment period (Day 1 to Day 43)
  Maximum concentration (Cmax) of TGRX-678 measured in plasma
Plasma AUC(0-t) | During Treatment period (Day 1 to Day 43)
  Area Under drug concentration-time curve (AUC) from time 0 to last measureable timepoint for TGRX-678 as measured in plasma
Plasma AUC(0-inf) | During Treatment period (Day 1 to Day 43)
  Area Under drug concentration-time curve from time 0 to infinity for TGRX-678 as measured in plasma
AUC(%Extrap) | During Treatment period (Day 1 to Day 43)
  Calculated percentage of Area under curve for AUC(0-inf) that is from last measurable timepoint ot infinity, calculated based on TGRX-678 plasma concentration over time curve.
Half Life (T1/2) | During Treatment period (Day 1 to Day 43)
  Time for TGRX-678 to decrease from maximum plasma concentration to half of maximum plasma concentration
Plasma volume of distribution (Vz/F) | During Treatment period (Day 1 to Day 43)
  Apparent volume of distribution of TGRX-678 in plasma
Plasma clearance (CL/F) | During Treatment period (Day 1 to Day 43)
  Apparent clearance of TGRX-678 in plasma

SECONDARY OUTCOMES:
Adverse Events (AE) | Starting from consent signing and until end of Treatment period (Day 1 to Day 43)
  To record adverse events to participants during study participation

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, MD, Principal Investigator — Nanjing Drug Tower Hospital
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No